CLINICAL TRIAL: NCT06425900
Title: Histologic and Liquid Chromatography Mass Spectrometry (LCMS) Evaluation of the Sebaceous Gland Changes Induced by Clascoterone Cream 1%
Brief Title: A Study to Assess Sebaceous Gland Changes and Constituents of Sebum (Skin Oil) Induced by Clascoterone 1% Cream in Acne Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCS-115-22
Record Dates: First submitted 2024-05-10; First posted 2024-05-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Winlevi (Clascoterone ) cream 1% (Experimental)
  Interventions: Drug: Winlevi (Clascoterone) cream 1%

INTERVENTIONS:
Drug: Winlevi (Clascoterone) cream 1% — Dosed twice daily (BID)

SUMMARY:
to compare facial sebaceous gland morphology after 3 months of clascoterone cream 1% treatment and to compare facial sebum constituents at baseline to facial sebum constituents after 3 months of clascoterone cream 1% treatment

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects age 18-35 years.
2. Subjects of all Fitzpatrick skin types.
3. Subjects with moderate facial acne and prominent pores indicating sebaceous gland activity.
4. Subjects with oily facial skin.
5. Subjects who agree to use only the study product and nothing else to the face.
6. Subject must possess no scars or tattoos or other confounding dermatologic conditions on the face in the preauricular biopsy sites on the left and right face.
7. Subjects agree not to introduce any new skin care products during the study.
8. No known medical conditions that, in the investigator's opinion, may interfere with study participation.
9. Subjects have signed an Informed Consent Form in compliance with 21CFR Part 50: "Protection of Human Subjects."
10. Subjects are dependable and able to follow directions and willing to comply with the schedule of visits.
11. Subjects in generally good physical and mental health.

Exclusion Criteria:

1. Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics.
2. Subjects who are not willing to use the assigned study product to their face as instructed.
3. Subjects who have used any topical prescription products on the face for 4 weeks prior to study entry.
4. Subjects who have used any OTC products on the face for 2 weeks.
5. Subjects with clinically significant unstable medical disorders.
6. Subjects who are unwilling or unable to comply with the requirements of the protocol.
7. Subjects who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
8. Subjects currently participating in any other clinical trial.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the histologic demonstration of reduced facial sebaceous gland size when comparing baseline to 3 months of clascoterone cream 1 % treatment. | Week 12

SECONDARY OUTCOMES:
The secondary efficacy endpoint is the changes in sebum composition when comparing baseline to 3 months of clascoterone cream 1 % treatment. | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States